CLINICAL TRIAL: NCT05106751
Title: A Randomized, Multicenter, Evaluator-Blinded, Active-Controlled, Parallel-Group Investigation to Evaluate the Performance and Safety of YVOIRE® Classic Plus Versus Comparator for Temporary Correction of Nasolabial Folds
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LG-HACL033
Record Dates: First submitted 2021-10-24; First posted 2021-11-04 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-08

CONDITIONS: Correction of Nasolabial Folds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YVOIRE Classic plus (Experimental)
  Interventions: Device: Hyaluronic acid dermal filler
- Restylane Lidocaine (Active Comparator)
  Interventions: Device: Hyaluronic acid dermal filler

INTERVENTIONS:
Device: Hyaluronic acid dermal filler — Hyaluronic acid dermal filler used for facial volume or wrinkle correction

SUMMARY:
A Study to Evaluate the Performance and Safety of YVOIRE Classic plus on NLF.

DETAILED DESCRIPTION:
This is a Randomized, Multicenter, Evaluator-Blinded, Active-Controlled, Parallel-Group Study to Evaluate the Performance and Safety of YVOIRE Classic plus Versus Comparator for Temporary Correction of Nasolabial Folds.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 21 years or above age.
* 2 or 3 of the 5-point (0-4) NLFRS (Nasolabial Fold Rating Scale).
* Agree to use proper contraception as guided in the protocol.
* Signed for Informed Consent.

Exclusion Criteria:

* have received permanent facial implants anywhere in the face or neck or planning during the investigation.
* have undergone facial plastic surgery of the lower face and nasolabial region within 12 weeks
* have undergone semi-permanent filler in lower face
* have undergone temporary dermal filler treatment in the lower two-thirds of face within 12 months
* Have undergone facial tissue augmentation or facial treatment with fat or botulinum injections in the lower two-thirds of face
* Have undergone mesotherapy or cosmetic procedures in face or neck within 6 months
* have used any over-the-counter anti-wrinkle products or prescription anti-wrinkle medicines for the nasolabial folds within 28 days

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Mean change on the Nasolabial Fold Rating Scale (NLFRS) from baseline to Week24. | 24 weeks from baseline
  To evaluate the performance of YVOIRE Classic plus on Nasolabial Fold 24 weeks after treatment, the mean change from baseline to 24 weeks will be measured using 5-point Nasolabial Fold Rating Scale (NLFRS). NLFRS Grades are 0 (None/Minimal), 1 (Mild), 2 (Moderate), 3 (Severe), and 4 (Extreme).
Responder rate calculated using Nasolabial Fold Rating Scale (NLFRS) for Nasolabial fold at Week 24. | 24 weeks from baseline
  To evaluate the performance of YVOIRE Classic plus on Nasolabial fold 24 weeks after treatment, the responder rate defined as ≥ 1-point improvement on the 5-point Nasolabial Fold Rating Scale (NLFRS) from baseline to 24 weeks will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- LG Chem investigational site 01, Darmstadt, Germany

IPD SHARING:
Plan to Share IPD: No